CLINICAL TRIAL: NCT00956813
Title: Phase III, Randomized, Placebo-controlled, Double-Blind Trial of Flaxseed for the Treatment of Hot Flashes
Brief Title: Flaxseed in Treating Postmenopausal Women With Hot Flashes Who Have a History of Breast Cancer or Other Cancer or Who Do Not Wish to Take Estrogen Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N08C7; NCCTG-N08C7; CDR0000644811 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01928 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Hot Flashes; Menopausal Symptoms; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: menopausal symptoms; hot flashes; breast cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral flaxseed in the form of a bar similar to a granola bar once daily.
  Interventions: Dietary Supplement: flaxseed
- Arm II (Placebo Comparator): Patients receive oral placebo bar once daily.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: flaxseed — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Estrogen can relieve the symptoms of menopause, but can also cause the growth of breast cancer cells. Flaxseed may reduce the number of hot flashes and improve mood and quality of life in postmenopausal women not receiving estrogen therapy.

PURPOSE: This randomized phase III trial is studying flaxseed to see how well it works in treating postmenopausal women with hot flashes who have a history of breast cancer or other cancer or who do not wish to take estrogen therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy of flaxseed on hot flash scores in women with a history of breast cancer or other cancer or in women who do not wish to take estrogen therapy for fear of increased risk of breast cancer as measured by a daily prospective hot flash diary.
* To evaluate the side effect profile of flaxseed in this population.
* To evaluate the effects of flaxseed on mood (per the Profile of Mood States) and broader menopausal symptoms (per the MENQOL), daily interference from hot flashes (per the HFRDIS), and perception of benefit (per Global Impression of Change).

OUTLINE: Patients are stratified according to age (18-49 years vs ≥ 50 years); treatment with tamoxifen citrate, selective estrogen receptor modulators, or aromatase inhibitors (yes vs no); duration of hot flashes (≤ 9 months vs > 9 months); and daily frequency of hot flashes (4-9 vs ≥ 10). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral flaxseed in the form of a bar similar to a granola bar once daily.
* Arm II: Patients receive oral placebo bar once daily. In both arms, treatment continues for 6-12 weeks. Patients in arm II may crossover to receive treatment as in arm I after 6 weeks.

Patients complete questionnaires (Hot Flash Diary, Side Effect Experience Questionnaire, Profile of Mood States, Hot Flash Related Daily Interference Scale, and Menopause Specific Quality of Life) at baseline and periodically during treatment. Patients are contacted by telephone at the end of weeks 2, 4, 5, and 7 to assess product tolerability, document compliance, encourage completion of questionnaires, and address problems.

ELIGIBILITY:
* Bothersome hot flashes, defined by their occurrence ≥ 28 times per week and of sufficient severity to make the patient desire therapeutic intervention

  * Presence of hot flashes for ≥ 1 month
* Meets 1 of the following criteria:

  * History of breast cancer or other cancer (currently without malignant disease)
  * No history of breast cancer and wishes to avoid estrogen due to a perceived increased risk of breast cancer
* Hormone receptor status not specified
* Postmenopausal as defined by 1 of the following*:

NOTE: *Women with ≥ 1 ovary but without a uterus should be deemed postmenopausal by either age > 55 OR a combination of estrogen within a postmenopausal range (per local lab) and follicle-stimulating hormone > 40 mIU/mL

* Absence of a period in the past 12 months
* Bilateral oophorectomy

  * ECOG performance status 0-1
  * Life expectancy ≥ 6 months
  * Able to complete questionnaire(s) alone or with assistance
  * No diabetes requiring oral or injectable antihyperglycemics
  * No hypotension
  * No history of allergic or other adverse reaction to flaxseed
  * No irritable bowel syndrome, colitis, Crohn disease, or any gastrointestinal condition where the patient should not consume and/or has an intolerance/allergies to seeds or nuts
  * At least 4 weeks since prior and no concurrent or planned androgens, estrogens, or progestational agents
* Tamoxifen, raloxifene, or aromatase inhibitors are allowed provided the patient has been on a constant dose for ≥ 4 weeks and is not expected to stop the medication during study treatment

  • At least 4 weeks since prior and no concurrent anti-cancer therapies of any kind
* Trastuzumab allowed

  * No concurrent treatment with other anti-cancer therapies of any kind except for trastuzumab or endocrine therapies
  * No concurrent (≤ 7 days prior to registration) or planned use of other agents for treating hot flashes (i.e., gabapentin, clonidine, antidepressants, estrogen treatment, megestrol acetate, or Bellergal)
* Stable dose of vitamin E (as a general vitamin supplement) allowed provided it is ≤ 800 IU/day, it was started > 30 days before study initiation, and is to be continued through study period
* Patients who have been using antidepressants for mood and have been on a stable dose for over a month and meet the eligibility criteria for hot flash frequency and duration are eligible

  • No concurrent anticoagulants or anti-platelets (1 mg of Coumadin for central line patency allowed)
* Aspirin allowed (≤ 81 mg)

  * No concurrent anti-hypertensives
  * No other concurrent herbal supplements for any reason, including soy and soy supplements (i.e., powders, pills, or milk)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (107):
- United States (107):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Drs. Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Pruthi S, Qin R, Terstreip SA, Liu H, Loprinzi CL, Shah TR, Tucker KF, Dakhil SR, Bury MJ, Carolla RL, Steen PD, Vuky J, Barton DL. A phase III, randomized, placebo-controlled, double-blind trial of flaxseed for the treatment of hot flashes: North Central Cancer Treatment Group N08C7. Menopause. 2012 Jan;19(1):48-53. doi: 10.1097/gme.0b013e318223b021. PMID 21900849
- [Result] Pruthi S, Qin R, Terstriep SA, et al.: The evaluation of flaxseed for hot flashes: results of a randomized, controlled trial, NCCTG study N08C7. [Abstract] J Clin Oncol 29 (Suppl 15): A-CRA9015, 2011.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One-hundred-five patients were randomized to each of the Flaxseed arm and the Placebo arm. After unblinding, all patients had the option of continuing Flaxseed treatment for 6 additional weeks to obtain longer term information about the effects of flaxseed for the management of hot flashes and to allow the placebo arm to try the flaxseed.
Groups:
- Flaxseed: Patients receive 1 Nutrigrad™ flaxseed bar containing 7.5 grams flaxseed, 410 mg lignans,once daily.
- Placebo: Patients Identical looking bar with same calorie and total fat content but without flaxseed or lignans once daily.
Period: Flaxseed and Placebo
Arm/Group | Flaxseed | Placebo
Started | 105 | 105
Completed | 97 | 100
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Ineligible | 3 | 1
Period: Continuation Phase
Arm/Group | Flaxseed | Placebo
Started | 80 | 0
Completed | 80 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that registered are included in baseline characteristics for the Flaxseed and Placebo Period. Patients who continued treatment during the Optional Continuation Period were a subset of the original 210 patients and are reported separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flaxseed | Placebo | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Customized [Count of Participants; unit: Participants] — Population: Patients that continued with the Optional Flaxseed Continuation Period were combined for baseline analysis.
  Participants
    Flaxseed and Placebo Period: <50 | 25 | 24 | 49
    Flaxseed and Placebo Period: >=50 | 80 | 81 | 161
    Optional Flaxseed Continuation: number analyzed (Participants) | 80 | 0 | 80
    Optional Flaxseed Continuation: <50 | 25 |  | 25
    Optional Flaxseed Continuation: >=50 | 55 |  | 55
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Patients that continued with the Optional Flaxseed Continuation Period were combined for baseline analysis.
  Participants
    Flaxseed and Placebo Period: Female | 105 | 105 | 210
    Flaxseed and Placebo Period: Male | 0 | 0 | 0
    Optional Flaxseed Continuation: number analyzed (Participants) | 80 | 0 | 80
    Optional Flaxseed Continuation: Female | 80 | 0 | 80
    Optional Flaxseed Continuation: Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 105 | 105 | 210

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of Flaxseed on Hot Flash Scores in Women as Measured by a Daily Prospective Hot Flash Diary.
Description: The intra-patient difference in hot flash activity between baseline (study week 1) and treatment termination (study week 7) is the primary endpoint. The hot flash activity will be measured by the weekly average hot flash score which is a composite entity of both frequency and severity of hot flashes.
  The hot flash severities are graded from 1 to 4, ranging from mild, to moderate, to severe to very severe. The daily hot flash score is computed by multiplying the mean grade of severity by the frequency during every 24 hour period. Therefore, a score of zero is the lowest possible score and can be interpreted as having no hot flashes. The average daily hot flash score during the baseline week was compared to the average daily value during week 7.
  The primary method of analysis will be the independent sample t-test to examine the change of weekly average hot flash score from baseline to treatment termination between flaxseed and placebo arms.
Time Frame: Baseline and 7 weeks
Population: Per protocol, the study was powered for 77 patients on each arm. With 20% over-accrual, the analysis began after 94 patients registered to each arm. 25 patients from Flaxseed were not used (4 cancel, 2 ineligible, 12 refused further treatment, 5 due to adverse events, 2 noncompliance). 17 from the placebo arm were not used (3,1,5,7,1 respective)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flaxseed | Placebo
Number analyzed (Participants) | 69 | 77
units on a scale | -4.9 (6.41) | -3.5 (6.47)
Statistical Analysis 1: Comparison: Flaxseed vs Placebo; Test type: Superiority or Other; p = 0.29, t-test, 2 sided

2. Secondary Outcome: Toxicity as Measured by CTCAE v3.0
Description: Frequency and severity of adverse events were reported by patients weekly evaluated through clinical assessment by NCI CTCAE v3.0. The number of patients reporting grade 3 or higher events are reported in this outcome measure. For a full list of all events, please refer to the Adverse Events section of this report.
Time Frame: Up to 7 weeks
Population: All patients treated during the Double-blinded period of the study were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Flaxseed | Placebo
Number analyzed (Participants) | 101 | 102
Participants
  Grade 3+ Adverse Event | 0 | 1
  Grade 4+ Adverse Event | 0 | 0

3. Secondary Outcome: Change of Mood as Measured by the Profile of Mood States (POMS)
Description: Profile of Mood States (POMS) was used to look at total mood disturbance as well as the subscales of tension-anxiety, fatigue-inertia, and vigor-activity. The POMS is a well known, well validated, reliable measure of psychological distress which includes 6 subscales of fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment. The entire scale can be scored to provide a measure of total mood disturbance. The measure contains adjectives related to mood which are scored from 0 (not at all) to 4 (extremely). Individual scores were converted to a 0-100 scale where 100 is best quality of life.
  The change of mood as measured by the POMS from baseline to treatment termination between flaxseed versus placebo arms was compared using Kruskal-Wallis test. The mean change in total score for each arm is reported.
Time Frame: Baseline and up to 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flaxseed | Placebo
Number analyzed (Participants) | 69 | 77
units on a scale | 6.6 (9.92) | 5.7 (9.41)
Statistical Analysis 1: Comparison: Flaxseed vs Placebo; Test type: Superiority or Other; p = 0.93, Kruskal-Wallis

4. Secondary Outcome: Change of Menopause Specific Quality of Life as Measured by the Menopause Specific Quality of Life (MENQOL)
Description: The change in quality of life as measured by the MENQOL from baseline to treatment termination between flaxseed versus placebo arms was evaluated. On a 0-6 scale, patients were asked to answer questions in in each of 4 domain scores (Vasomotor, Psychosocial, Physical, Sexual) Scores were converted to a 0-100 scale where 100 is best QOL. The change in score from baseline to end of treatment were analyzed separately for each domain. Here we report the mean change in score for each category.
Time Frame: Baseline and up to 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flaxseed | Placebo
Number analyzed (Participants) | 69 | 77
units on a scale
  Change in Vasomotor score | 22.5 (20.13) | 18.7 (22.04)
  Change in Psychosocial score | 9.9 (12.49) | 11.1 (15.02)
  Change in Physical Score | 9.3 (13.44) | 11.8 (15.19)
  Change in Sexual Score | 14.4 (18.27) | 14.4 (22.05)
Statistical Analysis 1: Comparison: Flaxseed vs Placebo; Testing the change in score from baseline to treatment completion for vasomotor-related questions in the MENQOL form; Test type: Superiority or Other; p = 0.19, Kruskal-Wallis
Statistical Analysis 2: Comparison: Flaxseed vs Placebo; Testing the change in score from baseline to treatment completion for Psychosocial-related questions in the MENQOL form; Test type: Superiority or Other; p = 0.78, Kruskal-Wallis
Statistical Analysis 3: Comparison: Flaxseed vs Placebo; Testing the change in score from baseline to treatment completion for Physical-related questions in the MENQOL form; Test type: Superiority or Other; p = 0.238, Kruskal-Wallis
Statistical Analysis 4: Comparison: Flaxseed vs Placebo; Testing the change in score from baseline to treatment completion for Sexually-related questions in the MENQOL form; Test type: Superiority or Other; p = 0.497, Kruskal-Wallis

5. Secondary Outcome: Change of Daily Interference as Measured by the Hot Flash Related Daily Interference Scale (HFRDIS)
Description: The change of daily interference as measured by the HFRDIS from baseline to treatment termination between flaxseed versus placebo arms was evaluated with an independent t-test for continuous data. On a 0-10 scale, patients were asked to describe how hot flashes interfered with 10 different aspects of their life (work, social activities, leisure activities, sleep, mood, concentration, relationships with others, sexuality, enjoyment of life and overall quality of life). Scores were converted to a 0-100 scale where 100 is best QOL.The HFRDIS total score was the average of the 10 individual questions. The change in total score from baseline to end of treatment was analyzed between the groups using a Kruskal-Wallace test.
Time Frame: Baseline and up to 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flaxseed | Placebo
Number analyzed (Participants) | 69 | 77
units on a scale | 13.9 (18.57) | 9.8 (19.65)
Statistical Analysis 1: Comparison: Flaxseed vs Placebo; Test type: Superiority or Other; p = 0.089, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: The Placebo and Flaxseed arm were the double-blinded first 7 weeks of treatment. After the 7 weeks of double-blinded treatment, patients were given the option of continuing treatment according to the Flaxseed arm for up to 6 additional weeks.
Description: Adverse events were assessed every week during treatment. All patients that began study treatment and were assessed at least once for adverse events were included in this analysis
Groups:
- Optional Continuation Period: After completing the Placebo/Flaxseed double-blind period, patients were allowed to continue with 1 Nutrigrad™ flaxseed bar containing 7.5 grams flaxseed, 410 mg lignans,once daily.
Arm/Group | Flaxseed | Placebo | Optional Continuation Period
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/102 | 0/76
Other Adverse Events (participants affected / at risk) | 61/101 | 71/102 | 32/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flaxseed (N=101) | Placebo (N=102) | Optional Continuation Period (N=76)
Abdominal distension (Gastrointestinal disorders) | 33 (53) | 30 (50) | 11 (21)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 11 (15) | 16 (19) | 6 (7)
Flatulence (Gastrointestinal disorders) | 45 (93) | 45 (79) | 27 (55)
Nausea (Gastrointestinal disorders) | 21 (29) | 16 (21) | 5 (8)
Vomiting (Gastrointestinal disorders) | 2 (3) | 6 (7) | 3 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (13) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 7 (13) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less